CLINICAL TRIAL: NCT02007486
Title: Pathophysiological Mechanisms of Activity-Related Dyspnea in Heart Failure: A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Other Study IDs: MCRDF 2013
Record Dates: First submitted 2013-11-28; First posted 2013-12-10 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Exercise; Dyspnea; Diaphragm electromyogram; Respiratory mechanics
MeSH Terms: conditions — Heart Failure; Motor Activity; Dyspnea | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Heart Failure: NYHA functional class I: Ambulatory and clinically-stable patients with New York Heart Association Functional Class I heart failure and a left ventricular ejection fraction (LVEF) on echocardiography of <45%.
  Interventions: Other: Cardiopulmonary Exercise Testing
- Heart Failure: NYHA functional class II: Ambulatory and clinically-stable patients with New York Heart Association Functional Class II heart failure and a left ventricular ejection fraction (LVEF) on echocardiography of <45%.
  Interventions: Other: Cardiopulmonary Exercise Testing
- Heart Failure: NYHA functional class III: Ambulatory and clinically-stable patients with New York Heart Association Functional Class III heart failure and a left ventricular ejection fraction (LVEF) on echocardiography of <45%.
  Interventions: Other: Cardiopulmonary Exercise Testing
- Healthy Control Subjects: Healthy, sedentary, non-smoking, age- and sex-matched control subjects.
  Interventions: Other: Cardiopulmonary Exercise Testing

INTERVENTIONS:
Other: Cardiopulmonary Exercise Testing — Symptom-limited incremental exercise testing (10 watts/min) on an electronically braked cycle ergometer

SUMMARY:
Dyspnea (breathlessness) on exertion is the most prevalent and distressing symptom of heart failure (HF). Nevertheless, the mechanisms of dyspnea in HF remain poorly understood. Thus, the general aim of this pilot study is to advance our understanding of the mechanisms of activity-related dyspnea in patients with HF. Studies will be performed in patients with mild, moderate and severe HF (n=24) as well as in healthy, age- and sex-matched control subjects (n=8). We will test the hypothesis that the increased prevalence and severity of activity-related dyspnea in HF reflects the interaction between an exaggerated drive to breathe and the inability of the respiratory system to meet this increased demand. Detailed physiological and perceptual responses to bicycle exercise will be examined and compared, first, between HF patients and healthy control subjects and, second, across patients with varying degrees of HF severity. The results from this preliminary study will be used to help design future studies in this patient population.

ELIGIBILITY:
Inclusion Criteria for Heart Failure Patients:

* Male or Female
* Greater than or equal to 40 years
* Greater than or equal to 6 month history of Heart Failure due to ischemic or idiopathic causes
* New York Heart Association Functional Class I (n=8), II (n=8) and III (n=8)
* Ambulatory
* Clinically Stable, as evidenced by no change in medication dosage or frequency of administration and no exacerbations or hospitalizations due to Heart Failure in the preceding 3-months
* Left Ventricular Ejection Fraction on echocardiography of less than or equal to 45% determined in the preceding 12-months.

Exclusion Criteria for Heart Failure Patients:

* Chronic obstructive lung disease and/or active disease other than Heart Failure (e.g., bronchial asthma; pulmonary arterial hypertension that is not considered secondary to left heart failure; peripheral artery disease; primary valvular disease; neurological, cognitive, neuromuscular, endocrine, kidney, metabolic and/or musculoskeletal disease)
* Unstable angina
* Intermittent claudication
* History of dangerous cardiac arrhythmias
* Myocardial infarction and/or stroke in the preceding 6-months
* Use of a pacemaker or cardiac resynchronization device
* Use of domiciliary oxygen and/or exercise-induced arterial oxyhemoglobin desaturation to <80% on room air
* Current and/or ex-smoker with a cigarette smoking history of greater than or equal to 10 pack years
* Body mass index less than 18.5 or greater than or equal to 35.0 kg/m2
* Use of antidepressant, opioid and/or anti-coagulant drugs in the preceding 4-weeks
* Evidence of periodic breathing (or oscillatory ventilation) on initial exercise testing
* Evidence of significant sleep-disordered breathing (i.e., apnea-hypopnea index >15 events/hour of sleep) based on overnight polysomnography performed within preceding 12-months.

Inclusion Criteria for Healthy Control Subjects:

* Male or Female
* Greater than or equal to 40 years
* Non-smoker

Exclusion Criteria for Healthy Control Subjects:

* History of cardiovascular, cerebrovascular, pulmonary, musculoskeletal, neuromuscular, renal, endocrine, metabolic, neurologic and/or cognitive disease/dysfunction.
* Evidence of exercise-induced myocardial ischemia on ECG
* Evidence of exercise-induced oxyhemoglobin desaturation to <80% on room air
* Taking regular medication(s)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory, male and female heart failure patients (n=24) will be recruited from the Heart Failure and Heart Transplant Centre of the Royal Victoria Hospital, McGill University Health Centre. Healthy, sedentary, non-smoking, asymptomatic, control subjects (n=8) will be recruited through advertisement in the Montréal and surrounding area
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Sensory intensity (Borg 0-10 scale) ratings of dyspnea at a standardized sub-maximal work rate during exercise | Patients will be followed until all study visits are complete, an expected average of 2 weeks

SECONDARY OUTCOMES:
Esophageal electrode catheter-derived measurements of the diaphragm EMG at a standardized sub-maximal work rate during exercise. | Patients will be followed until all study visits are complete, an expected average of 2 weeks
Power output (measured in watts) at the symptom-limited peak of incremental cycle ergometer exercise testing | Patients will be followed until all study visits are complete, an expected average of 2 weeks.
  The highest power output (measured in watts) that the study participants are able to sustain for greater than or equal to 30 seconds will be defined as the "symptom-limited peak power output" and used as a secondary outcome measure in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- McConnell Centre for Innovative Medicine, Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl